CLINICAL TRIAL: NCT02796157
Title: A Randomized Comparison of Clinical Outcomes Between Everolimus-eluting Bioresorbable Vascular Scaffold Versus Everolimus-eluting Metallic Stent in Long Coronary Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2016-0025
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease
Keywords: bioresorbable vascular scaffold, drug eluting stent, coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- absorb arm (Active Comparator): PCI with Absorb everolimus-eluting bioresorbable vascular scaffold
  Interventions: Device: PCI with Absorb everolimus-eluting bioresorbable vascular scaffold
- Xience arm (Experimental): PCI with Xience everolimus-eluting metallic stent
  Interventions: Device: PCI with Xience everolimus-eluting metallic stent

INTERVENTIONS:
Device: PCI with Absorb everolimus-eluting bioresorbable vascular scaffold — Patients allocated to this arm will undergone PCI with Absorb everolimus-eluting bioresorbable vascular scaffold. It will be allowed to used multiple stents for a long coronary lesion.
  Arms: absorb arm
Device: PCI with Xience everolimus-eluting metallic stent — Patients allocated to this arm will undergone PCI with Xience everolimus-eluting metallic stent. It will be allowed to used multiple stents for a long coronary lesion.
  Arms: Xience arm

SUMMARY:
PCI of diffuse long coronary lesions still remains challenging because of relatively high risk of in-stent restenosis and stent thrombosis compared to short coronary lesions. The purpose of the study is to compare an incidence of composite of major adverse cardiovascular events (MACEs) at 1 year between Absorb everolimus-eluting BVS and Xience EES after coronary intervention in long lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-85 years
* Patients with ischemic heart disease requiring PCI
* Significant coronary de novo lesion (stenosis >50% by quantitative angiographic analysis) requiring stent ≥28 mm in length based on angiographic estimation
* Reference vessel diameter of 2.5 to 3.75 mm by operator assessment

Exclusion Criteria:

* Acute myocardial infarction within 48 hours with unstable hemodynamics requiring pharmacologic or mechanical support
* Complex coronary morphology including left main disease and bifurcation lesion requiring two-stent technique
* Contraindication or hypersensitivity to anti-platelet agents or contrast media
* Treated with any metallic stent or BVS within 3 months at other vessel
* Cardiogenic shock
* Left ventricular ejection fraction <40%
* Pregnant women or women with potential childbearing
* Inability to follow the patient over the period of 1 year after enrollment, as assessed by the investigator
* Inability to understand or read the informed content

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 950 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite of major adverse cardiovascular events | 1 year after PCI
  Cardiac death, nonfatal myocardial infarction (MI), stent thrombosis and target-lesion revascularization (TLR)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Seo J, Ahn JM, Hong SJ, Kang DY, Hong SJ, Her AY, Kim YH, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Jang Y, Park SJ, Park DW, Hong MK. Bioresorbable Vascular Scaffolds Versus Drug-Eluting Stents for Diffuse Long Coronary Narrowings. Am J Cardiol. 2020 Jun 1;125(11):1624-1630. doi: 10.1016/j.amjcard.2020.02.031. Epub 2020 Mar 15. PMID 32279841